CLINICAL TRIAL: NCT02658071
Title: Measurement of Ocular Tensional Fluctuation by Triggerfish Lens Before and After Cataract Surgery in Patients With Exfoliative Glaucoma
Acronym: TRIGGERFISH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Sensimed AG (Industry)
Responsible Party: Sponsor
Other Study IDs: TRIGGERFISH (RB 15.063)
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Cataract; Exfoliative Glaucoma
Keywords: exfoliative glaucoma; cataract; ocular pressure
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is a very frequent disease in Brittany. In glaucoma the retinal ganglion cells and their axons slowly die with visible changes at the optic nerve head (cupping). Without early diagnosis and effective treatment or with delayed treatment decrease of visual acuity or blindness become.

In secondary pseudoexfoliation glaucoma grayish-white deposits of abnormal proteins are found on all surfaces of eye irrigated by the aqueous humor. The deposits of PEX material inside the trabecular meshwork decrease aqueous humour outflow and the intraocular pression raise. The exfoliation material is found on the surface of the lens capsule with frequent developement of nuclear cataract . After cataract surgery the intra ocular pressure (IOP) decrease.

Some recent study have found decreasing ocular volume variation associated to IOP fluctuation in night after cataract surgery in normal pressure glaucoma patients. In our study we want see if it's the same thing in pseudoexfoliation glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Exfoliative glaucoma
* Patient who need cataract surgery
* Patient agree with study

Exclusion Criteria:

* Monophtalm patient
* Patient with bleb after glaucoma surgery
* Terminal glaucoma
* Herpes
* One year control impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with exfoliative glaucoma and cataract
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-03-15 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
Measurement of ocular tensional fluctuation by Triggerfish lens before and after cataract surgery in patients with exfoliative glaucoma. | During 24H00 before and after cataract surgery
  Variation of ocular volume

CONTACTS AND LOCATIONS:
Overall Officials: Catherine COCHARD, Dr, Principal Investigator — University Hospital of Brest
Locations (1):
- CHRU de Brest, Brest, France